CLINICAL TRIAL: NCT00603018
Title: PET Imaging of Dopaminergic Transmission and Serotonin Markers in Anorexia Nervosa
Brief Title: PET Imaging Study of Recovered Anorexics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Walter Kaye, MD/Director, Eating Disorders Program Professor,, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO06110005
Record Dates: First submitted 2007-10-16; First posted 2008-01-28 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Anorexia Nervosa
Keywords: eating disorders; anorexia nervosa; anorexia; PET; brain imaging; serotonin; fMRI; Prozac; fluoxetine
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Anorexia | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Annorexia nervosa (Experimental): Participants recovered from anorexia nervosa before and after administration of fluoxetine
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — 8 weeks of fluoxetine(2.5mg,5mg,10mg,20mg,30mg,40mg,40mg,40mg)each week per day.
  Other Names: Prozac

SUMMARY:
Several studies in the past suggest that individuals who have or had anorexia nervosa may have alterations in brain serotonin. Serotonin seems to play an important role in regulating anxiety, mood, and other symptoms found in anorexia nervosa. We will be using a technology called Positron Emission Tomography (PET), which is a method used to take pictures of the body, in this case, the brain. Study participants will undergo two baseline PET scans on the first day of the study. The women who have recovered from anorexia will then be given a medication called fluoxetine (also know as Prozac) to take for 8 weeks. At the end of the 8th week, they will return for a third PET scan. By comparing the brain scans, before and after fluoxetine treatment, we can understand more about how treatment with fluoxetine affects the serotonin receptors in the brain. We will be comparing brain serotonin system in women who have recovered from anorexia before and after medication in order to gain a better understanding of changes in the serotonin system associated with eating disorders. This study may help shed light on how to make fluoxetine a more effective treatment for anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Recovered from Anorexia Nervosa
* Not taking medication for emotional problems
* Regular menstrual cycle

Exclusion Criteria:

* Women who are pregnant or nursing
* Psychoactive medications in the past 30 days
* Neurological disorders.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kaye, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/15992780?ordinalpos=40&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Recovered From Anorexia Before + After Fluoxetine: Participants recovered from anorexia
  Fluoxetine: before 8 weeks of fluoxetine(2.5mg,5mg,10mg,20mg,30mg,40mg,40mg,40mg)each week per day.
Period: Overall Study
Arm/Group | Participants Recovered From Anorexia Before + After Fluoxetine
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 1/Recovered Anorevia: Recovered anorexia
  Fluoxetine: 8 weeks of fluoxetine(2.5mg,5mg,10mg,20mg,30mg,40mg,40mg,40mg)each week per day.
Arm/Group | 1/Recovered Anorevia
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Serotonin Receptor 1A Binding Potential In Regions of Interest (ROI) Accounting for Binding Potential in a Region Without Serotonin 1A Receptors
Description: We used PET and [11C]WAY to assess 5-HT1A binding potential (BP) = [11C]WAY 100635 BP = Distribution Volume (DV)ROI-DVcerebellum in striatal regions; subcortical regions including insula, medial temporal lobe, amygdala, hippocampus, midbrain, parahippocampal gyrus; and the neocortical regions (i.e., anterior cingulate cortex). Analysis of the PET data was performed using the Logan graphical method (Logan et al. 2001) with the cerebellum as a reference region for non-displaceable uptake. 23 REC AN were studied. The Binding Potential (BP) was calculated as followed: BPP = fP Bavail/KD = VT-VND;(Abbrev.: BPP = In vivo binding potential; fP = free fraction in plasma; Bavail = Density of receptors available to bind radioligand in vivo; KD = Dissociation Constant; V = Volumes of Distribution expressed relative to total plasma ligand concentration; T = Total radioligand in tissue; ND = Nondisplaceable tissue uptake; see Innis et al. 2007); Units: mL cm -3
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mL/cm^3
Groups:
- 1/Recovered Anorexia Before 8 Weeks of Treatment: 1/Recovered anorexia before 8 weeks of treatment
  Baseline
- 1/Recovered Anorexia After 8 Weeks of Treatment: 1/Recovered anorexia after 8 weeks of treatment
  Fluoxetine: 8 weeks of fluoxetine(2.5mg,5mg,10mg,20mg,30mg,40mg,40mg,40mg)each week per day.
Arm/Group | 1/Recovered Anorexia Before 8 Weeks of Treatment | 1/Recovered Anorexia After 8 Weeks of Treatment
Number analyzed (Participants) | 23 | 23
mL/cm^3
  insula | 5.97 (1.43) | 5.89 (2.17)
  medial temporal lobe | 6.66 (2.14) | 6.91 (2.62)
  amygdala | 5.91 (2.85) | 6.29 (3.17)
  hippocampus | 9.08 (3.98) | 9.92 (4.75)
  midbrain | 0.37 (.16) | .58 (.36)
  anterior cingulate cortex | 3.83 (1.14) | 4.12 (1.73)
  parahippocampal gyrus | 6.08 (1.57) | 6.05 (1.79)

ADVERSE EVENTS:
Groups:
- 1/Recovered Anorexia: Recovered anorexia
  Fluoxetine: 8 weeks of fluoxetine(2.5mg,5mg,10mg,20mg,30mg,40mg,40mg,40mg)each week per day.
Arm/Group | 1/Recovered Anorexia
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes